CLINICAL TRIAL: NCT03349853
Title: Description of the Use of Subcutaneous Acetaminophen in Palliative Care Unit
Brief Title: Description of the Use of Subcutaneous Acetaminophen in Palliative Care Unit in France: Descriptive Questionnaire Survey
Acronym: EnPasc
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-04Obs-CHRMT
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Pain
Keywords: Palliative care; Acetaminophen; Subcutaneous route; Pain treatment
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acetaminophen is a drug commonly used in palliative care unit, for its antalgic and antipyretic effects. Several administration routes are possible but the use of the sub-cutaneous route is actually not supported by recommandations.

ELIGIBILITY:
Inclusion Criteria:

* doctors responsible for palliative care unit in France

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: doctors responsible for palliative care unit in France
Sampling Method: Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2016-06-18 (Actual); Study Completion 2016-06-18 (Actual)

PRIMARY OUTCOMES:
knowledge about the use of subcutaneous acetaminophen in palliative care unit. | day 1
  questionnaire